CLINICAL TRIAL: NCT02257502
Title: Phase II Study Evaluating the Efficacy of Aflibercept for the Treatment of Iodiopathic Choroidal Neovascularization in Young Patients
Brief Title: Study Evaluating the Efficacy of Aflibercept for the Treatment of NVCI in Young Patients
Acronym: INTUITION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013.839; 2013-005081-19 (EudraCT Number)
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Idiopathic Choroidal Neovascularization
Keywords: aflibercept; iodiopathic choroidal neovascularization; young patient
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- aflibercept (Experimental): intravitreal injection of aflibercept (EYLEA)
  Interventions: Drug: aflibercept

INTERVENTIONS:
Drug: aflibercept — The patients are followed on a monthly basis until 52 weeks. Intravitreal injections of aflibercept at a dosage of 2 mg are initiated with a TAE regimen until 20 weeks (3 mandatory injections at inclusion, week 8 and 20 with reinjection at week 4, 12 and 16 only in case of CNV activity). Then, a PRN regimen is considered until 52 weeks (reinjection in case of CNV activity). Therefore, each patient receives between 3 and 13 injections in the whole study.

SUMMARY:
After myopia, the second etiology of choroidal neovascularization (CNV) in young adults (<50 years old) is idiopathic choroidal neovascularization (ICNV) whose etiology remains unknown. This is a rare and severe disease, which can lead to blindness.

ICNV is treated at the moment with off-label anti-VEGF (Vascular Endothelial Growth Factor) therapy and could also benefit from aflibercept (EYLEA), a new anti-VEGF currently indicated in Age-related Macular Degeneration (AMD). Case reports suggest that such patients would not need as many injections as in AMD.

INTUITION is an open-label, single arm, prospective, multicenter, phase II study. The main objective is to demonstrate the effectiveness in clinical terms after 52 weeks of treatment with aflibercept on the visual acuity of patients affected by ICNV. A specific dosage regimen is designed to achieve maximum efficiency. The patients are followed on a monthly basis until 52 weeks. Intravitreal injections of aflibercept are initiated with a Treat & Extend (TAE) regimen until 20 weeks (3 mandatory injections with reinjection only in case of CNV activity). Then, a pro re nata (PRN) regimen is considered until 52 weeks (reinjection in case of CNV activity).

ELIGIBILITY:
Inclusion Criteria:

* 18 < Age < 50 years old
* Patient who give voluntary signed informed consent
* Patient affiliated with the French universal health care system or similar
* Patient with ICNV with active primary subfoveal, retrofoveal or juxtafoveal lesions that affect the fovea as evidenced by angiography (fluorescein and/or indocyanin green) and/or SD-OCT in the studied eye
* Patient willing, committed and able to return for all clinic visits and complete all study-related procedures

Exclusion Criteria:

* Pregnant women
* Sexually active men or women of childbearing potential who are unwilling to practice adequate contraception during the study
* Patient who is protected adults according to the terms of the law (French public health laws)
* Involvement in another clinical trial (studied eye and/or the other eye)
* Patient with non-ICNV, especially:

  * AMD
  * High myopia defined as refraction ≥ - 6 diopters
* Other curative treatment of ICNV in the studied eye during the last 3 months before the first intravitreal injection: anti-VEGF therapy, juxta- or extra-foveal macular laser, photodynamic therapy, surgery, external radiotherapy, transpupillary thermotherapy ...
* Medical history of retrofoveal focal macular laser photocoagulation in the studied eye
* Subretinal haemorrhage reaching the fovea centre, with a size > 50% of the lesion area
* Fibrosis or retrofoveal retinal atrophy in the studied eye
* Retinal pigment epithelial tear reaching the macula in the studied eye
* Medical history of intravitreal medical device in the studied eye
* Medical history of auto-immune or idiopathic uveitis
* Proved diabetic retinopathy
* Intra-ocular pressure ≥ 25 mmHg despite two topical hypotonic treatments
* Aphakia or lack of lens capsule (not removed by YAG laser) in the studied eye
* Arterial hypertension that is not controlled by an appropriate treatment
* Previous or actual treatment with systemic administration of anti-VEGF therapy
* Known hypersensitivity to aflibercept, or another drug composite of the medicinal product used; allergy to fluorescein, indocyanin green, anaesthetic eye drops
* Active or suspected ocular or peri-ocular infection
* Serious active intra-ocular inflammation in the studied eye
* Medical history of intra-ocular surgery within 28 days before the first injection in the studied eye
* Any illness or ocular condition that would require an intra-ocular surgery in the studied eye within 12 months after the inclusion
* Follow up not possible during 12 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-07-06 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
Mean change in best-corrected visual acuity (BCVA) expressed as number of letters gained or lost measured with Early Treatment Diabetic Retinopathy Study (ETDRS) scale from baseline to week 52 | 52 weeks
  BCVA is measured on the ETDRS scale at an initial distance of 4 meters

SECONDARY OUTCOMES:
Mean change in BCVA expressed as number of letters gained or lost measured with ETDRS scale from baseline to week 24 | 24 weeks
Percentage of patients with a <15-letter loss in BCVA measured with ETDRS scale from baseline to week 24 | 24 weeks
Percentage of patients with a <15-letter loss in BCVA measured with ETDRS scale from baseline to week 52 | 52 weeks
Mean number of injections per patient during the TAE regimen (until week 20) | 20 weeks
Mean time to reinjection after TAE regimen (i.e. after the 3rd mandatory injection at week 20) | 32 weeks
Mean total number of injections per patient during the study | 52 weeks
Mean change in central retinal thickness (CRT) in micrometers measured with Spectral Domain - Optical Coherence Tomography (SD-OCT) from baseline to week 24 | 24 weeks
Mean change in CRT in micrometers measured with SD-OCT from baseline to week 52 | 52 weeks
Mean change in neovascular lesion size and morphology measured with fluorescein and/or indocyanin green angiography from baseline to week 52 | 52 weeks
Side-effects observed during the study | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Laurent KODJIKIAN, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon - Hôpital de la Croix-Rousse, Lyon, France

REFERENCES:
- [Result] Kodjikian L, Tadayoni R, Souied EH, Baillif S, Milazzo S, Dumas S, Uzzan J, Bernard L, Decullier E, Huot L, Mathis T. EFFICACY AND SAFETY OF AFLIBERCEPT FOR THE TREATMENT OF IDIOPATHIC CHOROIDAL NEOVASCULARIZATION IN YOUNG PATIENTS: The INTUITION Study. Retina. 2022 Feb 1;42(2):290-297. doi: 10.1097/IAE.0000000000003310. PMID 34620799